CLINICAL TRIAL: NCT02848157
Title: Effects of Dexmedetomidine as Adjunct to Pudendal Block for Pediatric Penile Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2016-0379
Record Dates: First submitted 2016-07-05; First posted 2016-07-28 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Elective Penile Surgeries; Hypospadias; Urethral Fistula or Stricture After Hypospadias Repair; Penile Curvature
Keywords: dexmedetomidine; pudendal block; hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DR (Experimental): dexmedetomidine 0.3mcg/kg and 0.25% ropivacaine 0.3ml/kg
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine
- PR (Placebo Comparator): 0.25% ropivacaine 0.3ml/kg
  Interventions: Drug: plain ropivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients are put in lithotomy position. Two separate injection points are marked at 3 and 9 o'clock, about 2 to 2.5 cm from the center of anus. After aseptic preparation, a nerve stimulator needle advanced 1.5 to 3.5 cm perpendicular to the skin, and stimulation current is 2.5 to 5 mA. The unilateral contraction of anal sphincter means the inferior anal nerve stimulation. After reducing the current to 0.5 mA, the needle is then moved deeper until an up-and-down penile movement is observed. This is stimulation of the perineal branch of the pudendal nerve. Prepared drug (0.25% ropivacaine and 0.3 mcg/kg dexmedetomidine in the experimental group, and equivalent doses of ropivacaine and normal saline in the control group) is injected in half and half bilaterally.
  Arms: DR
Drug: plain ropivacaine — ropivacaine and normal saline equivalent doses of dexmedetomidine
  Arms: PR
Drug: Ropivacaine
  Arms: DR

SUMMARY:
Caudal block is often performed to relieve postoperative pain in pediatric urological surgery. Recently, pudendal block is also used in penile surgery and it has advantage because of less side effects such as transient weakness of low extremities, but limited to use in penile surgery. Local anesthesia is a single shot injection, so additional analgesic drugs is required when the effect of local anesthetics are disappeared. Dexmedetomidine, an alpha adrenergic agonist, is commonly used in pediatric sedation. It has analgesic effect and potentiates the effect of local anesthetics. There are many studies about the potentiation of the effect of local anesthetics when added to dexmedetomidine in adults, it has been limited in pediatrics. Recent study said that local anesthetics with dexmedetomidine had prolonged duration of analgesia in caudal block, also in ilioinguinal block. Thus it is expected to have a prolonged effect when investigators use dexmedetomidine in pediatrics as well as adults.

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged between 6 months and 6 years in elective penile surgeries (hypospadias, urethral fistula or stricture after hypospadias repair, penile curvature)
2. American Society of Anesthesiologists (ASA) class I, II

Exclusion Criteria:

1. Coagulopathy
2. allergy to local anesthetics
3. meatal island onlay proximal transverse island flap (MIOPTI) (more than 4 h for the surgery)
4. illiteracy, foreigner

Max Age: 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
1st analgesic request time | until 24 hours after surgery
  time to first rescue medication, assessed up to 24 h (time frame: from the administration of the pudendal block to the first registration of a FLACC≥4) (FLACC: face, legs, activity, cry, consolability)

SECONDARY OUTCOMES:
Postoperative pain evaluated by the FLACC scale | The time of arrival in the recovery room, 10, 20, 30 min after arrival of the recovery room, and 4, 8, 12, 24 h after the surgery.
  Postoperative pain is evaluated by the FLACC scale
Emergence delirium evaluated by the pediatric anesthesia emergence delirium scale | The time of arrival in the recovery room, 10, 20, 30 min after arrival of the recovery room, and through the time of discharge from the PACU, an average of 30 minutes
  emergence delirium is evaluated by the pediatric anesthesia emergence delirium scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No